CLINICAL TRIAL: NCT06077552
Title: Effect of Pyramidal Training on Selected Risk Factors of Atherosclerosis in Women With Central Obesity
Brief Title: Effect of Pyramidal Training on Selected Risk Factors of Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004666
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Atherosclerosis
Keywords: obesity; risk factor; lipid profile
MeSH Terms: conditions — Obesity; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): pyramidal training by treadmill for 40 minutes per session three sessions per week for eight weeks in addition to the diet health advises.
  Interventions: Other: pyramidal training by treadmill
- control group (No Intervention): receive diet health advises.

INTERVENTIONS:
Other: pyramidal training by treadmill — pyramidal training by treadmill for 40 minutes per session three sessions per week for eight weeks in addition to the diet health advises
  Arms: experimental group

SUMMARY:
The study will be conducted on fifty women with central obesity. Their ages will be from 30-40 years old. They will be selected from Al Hayat specialized Hospital in Cairo, Egypt and The participants will be randomly assigned into two equal groups:

Group (A): study group, 25 participants will receive pyramidal training by treadmill for 40 minutes per session three sessions per week for eight weeks in addition to the diet health advices.

Group (B): Control group, 25 participants will receive diet health advices. The subjects will be selected from El Haya specialized Hospital, Cairo.

DETAILED DESCRIPTION:
The study will be conducted on fifty women with central obesity. Their ages will be from 30-40 years old. They will be selected from Al Hayat specialized Hospital in Cairo, Egypt and The participants will be randomly assigned into two equal groups:

Group (A): study group, 25 participants will receive pyramidal training by treadmill for 40 minutes per session three sessions per week for eight weeks in addition to the diet health advices.

Group (B): Control group, 25 participants will receive diet health advices. The subjects will be selected from El Haya specialized Hospital, Cairo. Before starting the procedure the participants target heart rate (THR) will be calculated from Karvonen formula as follow: target heart rate (THR) = maximum heart rate (HRmax) - resting heart rate × intensity + resting heart rate(RHR)(Yabe et al.,2021).

The formula 208-0.7•age yield more precise estimates of HRmax over a wide age range (Nes et al., 2013).

After calculating THR, the study group participants will be on a pyramidal training program of incremental and decremental levels as follow:

The course of the program will be 2 sets of pyramidal training with 10 minutes for rest between them. each set will be 5 levels of incremental and 5 levels of decremental aerobic exercise and each level 2 minutes on a treadmill. All these levels will be ranked according to a percentage from the THR; the ranking will be as follow:

1. Level one: will be set as a 20% walking of Karvonen formula.
2. Level two: will be set as a 30% running of Karvonen formula.
3. Level three: will be set as a 50%running of Karvonen formula.
4. Level four: will be set as a 70% running of Karvonen formula.
5. Level five: will be set as a 80% running of Karvonen formula The whole program will be 40 minutes with warm up and cool down 5 minutes of stretch exercise for each. Participants will be asked to get on the treadmill and start the program, the therapist is monitoring the heart rate by using a pulse oximeter, and when the participants reach targeted percent of Karvonen formula, the therapist set the treadmill by increasing the speed to enter or start the up next level till reaching the highest level then start the decremental phase of the pyramidal training. The therapist shifts between the level by time or targeted percent of Karvonen formula which comes first.

ELIGIBILITY:
Inclusion Criteria:

* 1) Fifty women with central obesity. 2) Waist circumference > 88 cm. 3) Their age will be ranged from 30-40years old. 4) Body mass index (BMI) from 30 to 34.9 kg/m2. 5) High normal or abnormal lipid profile (total cholesterol > 200 mg/dl, HDL< 35 mg/dl, or triglycerides >150 mg/dl) and atherogenic index of plasma (AIP) ranges 0.11-0.21 6) HOMA-IR > 2.9 7) They are clinically and medically stable. 8) All participants are sedentary activity level according to physical activity index.

Exclusion Criteria:

* 1) Participants with musculoskeletal problems (e.g., Sever osteoarthritis or difficulties in ambulation).

  2) Participants with uncontrolled pulmonary disease. (e.g., Exaggerated chronic obstructive pulmonary disease, acute asthma).

  3) Any participants who missed more than two weeks of the program or want to terminate the program.

  4) Participants with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure.

  5) The participants have hearing impairment or mental disorders. 6) Implanted pacemaker. 7) Diabetes and hypertension.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
atherogenic index of plasma | 8 weeks
  blood analysis

SECONDARY OUTCOMES:
Waist circumference | 8 weeks
  tape measurement
Body mass index | 8 weeks
  measurement weight on height
lipid profile | 8 weeks
  blood analysis
insulin resistance | 8 weeks
  homeostatic model assessment for insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Marwa elsayed, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
journal publishing article
Supporting Information: Study Protocol
Time Frame: after 4 years of publishing
Access Criteria: publishing journal web site